CLINICAL TRIAL: NCT00628095
Title: A PHASE 2A, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL-GROUP STUDY OF CE-224,535, AN ANTAGONIST OF THE P2X7 RECEPTOR, IN THE TREATMENT OF THE SIGNS AND SYMPTOMS OF RHEUMATOID ARTHRITIS IN SUBJECTS WHO ARE INADEQUATELY CONTROLLED ON METHOTREXATE
Brief Title: Study of CE-224,535 A Twice Daily Pill To Control Rheumatoid Arthritis In Patients Who Have Not Totally Improved With Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A6341009; 2008-000327-25 (EudraCT Number)
Record Dates: First submitted 2008-02-25; First posted 2008-03-04 (Estimated); Results first posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Arthritis, Rheumatoid
Keywords: rheumatoid arthritis DMARD methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — CE 224,535

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: CE-224,535
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CE-224,535 — 500 mg po BID
  Arms: Active
Drug: Placebo — no active ingredient
  Arms: Placebo

SUMMARY:
CE-224,535 is known to block a chemical that acts as a gateway to some of your immune cells. Blocking this gateway prevents the cells from pushing out 2 chemicals called IL-1 and IL-18 that are known to cause some of the inflammation seen in rheumatoid arthritis. It is hoped that taking this drug will reduce the symptoms of rheumatoid arthritis

ELIGIBILITY:
Inclusion Criteria:

* Active rheumatoid arthritis
* Incomplete response to methotrexate

Exclusion Criteria:

* Must not be on biologic therapies
* No recent infections

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-04-07 (Actual); Primary Completion 2009-02-04 (Actual); Study Completion 2009-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- United States (14):
  - Arizona Arthritis & Rheumatology Associates, P.C., Mesa, Arizona
  - Omega Research Consultants LLC, DeBary, Florida
  - Florida Arthritis Center, Lake Mary, Florida
  - Tampa Medical Group, PA, Tampa, Florida
  - American Health Network, Avon, Indiana
  - Best Clinical Trials, LLC (Administrative Only), New Orleans, Louisiana
  - George Stanley Walker, MD, New Orleans, Louisiana
  - Majid Abdul Jawad, MD, New Orleans, Louisiana
  - The Arthritis and Osteoporosis Center of Maryland, Frederick, Maryland
  - University Physicians, Columbia, Missouri
  - University of Missouri-Columbia, Columbia, Missouri
  - Arthritis Center of Reno, Reno, Nevada
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Arthritis Northwest, Spokane, Washington
- Clínica Santa María, Sección Reumatología, Providencia, Santiago, RM, Chile
- Czechia (3):
  - Revmatologicka ambulance, Česká Lípa
  - Revmatologicky ustav, Prague
  - Revmatologicka ambulance, Prague
- Investigadores Clinicos Asociados, México, D.F., Mexico
- Poland (3):
  - Krakowskie Centrum Medyczne NZOZ, Krakow
  - Zaklad Reumatologii i Immunologii Klinicznej, Poznan
  - Oddzial Reumatologiczno-Rehabilitacyjny IIR Ortopedyczno-Rehabilitacyjny, Poznan
- South Korea (2):
  - Inha University Hospital, Medicine/Rheumatology, Incheon
  - Pusan National University Hospital, Rheumatology, Internal Medicine, Pusan
- Spain (3):
  - Hospital Nuestra Señora de La Esperanza, Santiago de Compostela, A Coruña
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital General Universitario Gregorio Marañon, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Stock TC, Bloom BJ, Wei N, Ishaq S, Park W, Wang X, Gupta P, Mebus CA. Efficacy and safety of CE-224,535, an antagonist of P2X7 receptor, in treatment of patients with rheumatoid arthritis inadequately controlled by methotrexate. J Rheumatol. 2012 Apr;39(4):720-7. doi: 10.3899/jrheum.110874. Epub 2012 Mar 1. PMID 22382341
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6341009&StudyName=Study%20of%20CE-224%2C535%20A%20Twice%20Daily%20Pill%20To%20Control%20Rheumatoid%20Arthritis%20In%20Patients%20Who%20Have%20Not%20Totally%20Improved%20With%20Methotrexate

RESULTS

PARTICIPANT FLOW:
Groups:
- CE-224,535: CE-224,535 500 milligram (mg) tablet orally twice daily for 12 weeks.
- Placebo: Placebo tablet matched to CE-224,535 500 mg tablet orally twice daily for 12 weeks.
Period: Overall Study
Arm/Group | CE-224,535 | Placebo
Started | 53 | 47
Completed | 46 | 40
Not Completed | 7 | 7
Not completed — Adverse Event | 5 | 3
Not completed — Lack of Efficacy | 0 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo tablet matched to CE-224,535 500 milligram (mg) tablet orally twice daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | CE-224,535 | Placebo | Total
Number analyzed (Participants) | 53 | 47 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (10.8) | 53.1 (11.6) | 53.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 88
  Male | 9 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With American College of Rheumatology 20% (ACR20) Response at Week 12
Description: ACR20 response: compared to baseline, greater than or equal to (>=) 20 percent (%) improvement in tender joint count; >= 20% improvement in swollen joint count; and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 12
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of the randomized study medication. Last observation carried forward (LOCF) was used to impute missing ACR components before computing ACR20 response.
Measure: Number; unit: Percentage of participants
Arm/Group | CE-224,535 | Placebo
Number analyzed (Participants) | 53 | 47
Percentage of participants | 33.96 | 36.17
Statistical Analysis 1: Comparison: CE-224,535 vs Placebo; Treatment effect was estimated by the difference of percentages between the treatment groups, and tested using the normal approximation method; Test type: Superiority or Other; p = 0.591, Normal Approximation method; No adjustments for multiple comparisons were performed; Percent difference = -0.0221, 90% CI 2-sided [-0.17 to 0.13] — Power of 80% and a Type I error at 0.10 in a 1-sided test was calculated. Null hypothesis stated that there was no difference between the CE-224,535 and placebo arm groups, on the percentage of ACR 20 responders at Week 12

2. Secondary Outcome: Percentage of Participants With American College of Rheumatology 20% (ACR20) Response at Week 2, 4 and 8
Description: ACR20 response: compared to baseline, >=20% improvement in tender joint count; >= 20% improvement in swollen joint count; and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 2, 4, 8
Population: FAS included all randomized participants who received at least 1 dose of the randomized study medication. LOCF was used to impute missing ACR components before computing ACR20 response.
Measure: Number; unit: Percentage of participants
Arm/Group | CE-224,535 | Placebo
Number analyzed (Participants) | 53 | 47
Percentage of participants
  Week 2 | 13.21 | 25.53
  Week 4 | 32.08 | 38.30
  Week 8 | 30.19 | 29.79
Statistical Analysis 1: Comparison: CE-224,535 vs Placebo; Week 2: Treatment effect was estimated by the difference of percentages between the treatment groups, and tested using the normal approximation method; Test type: Superiority or Other; p = 0.941, Normal Approximation method; Percent difference = -0.1232, 80% CI 2-sided [-0.22 to -0.02]
Statistical Analysis 2: Comparison: CE-224,535 vs Placebo; Week 4: Treatment effect was estimated by the difference of percentages between the treatment groups, and tested using the normal approximation method; Test type: Superiority or Other; p = 0.742, Normal Approximation method; Percent difference = -0.0622, 80% CI 2-sided [-0.18 to 0.05]
Statistical Analysis 3: Comparison: CE-224,535 vs Placebo; Week 8: Treatment effect was estimated by the difference of percentages between the treatment groups, and tested using the normal approximation method; Test type: Superiority or Other; p = 0.482, Normal Approximation method; Percent difference = 0.0040, 80% CI 2-sided [-0.11 to 0.12]

3. Secondary Outcome: Percentage of Participants With American College of Rheumatology 50% (ACR50) Response
Description: ACR50 response: compared to baseline, >=50% improvement in tender joint count; >= 50% improvement in swollen joint count; and >= 50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 2, 4, 8, 12
Population: FAS included all randomized participants who received at least 1 dose of the randomized study medication. LOCF was used to impute missing ACR components before computing ACR50 response.
Measure: Number; unit: Percentage of participants
Arm/Group | CE-224,535 | Placebo
Number analyzed (Participants) | 53 | 47
Percentage of participants
  Week 2 | 5.66 | 6.38
  Week 4 | 7.55 | 8.51
  Week 8 | 13.21 | 12.77
  Week 12 | 11.32 | 17.02
Statistical Analysis 1: Comparison: CE-224,535 vs Placebo; Week 2: Treatment effect was estimated by the difference of percentages between the treatment groups, and tested using the Barnard exact test; Test type: Superiority or Other; p = 0.989, Barnard exact test; Percent difference = -0.0072, 80% CI 2-sided [-0.08 to 0.06]
Statistical Analysis 2: Comparison: CE-224,535 vs Placebo; Week 4: Treatment effect was estimated by the difference of percentages between the treatment groups, and tested using the Barnard exact test; Test type: Superiority or Other; p = 0.957, Barnard exact test; Percent difference = -0.0096, 80% CI 2-sided [-0.08 to 0.07]
Statistical Analysis 3: Comparison: CE-224,535 vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.473, Normal Approximation method; Percent difference = 0.0044, 80% CI 2-sided [-0.08 to 0.09]
Statistical Analysis 4: Comparison: CE-224,535 vs Placebo; Week 12: Treatment effect was estimated by the difference of percentages between the treatment groups, and tested using the normal approximation method; Test type: Superiority or Other; p = 0.793, Normal Approximation method; Percent difference = -0.0570, 80% CI 2-sided [-0.15 to 0.03]

4. Secondary Outcome: Percentage of Participants With American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response: compared to baseline, >=70% improvement in tender joint count; >= 70% improvement in swollen joint count; and >= 70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 2, 4, 8, 12
Population: FAS included all randomized participants who received at least 1 dose of the randomized study medication. LOCF was used to impute missing ACR components before computing ACR70 response.
Measure: Number; unit: Percentage of participants
Arm/Group | CE-224,535 | Placebo
Number analyzed (Participants) | 53 | 47
Percentage of participants
  Week 2 | 3.77 | 0.00
  Week 4 | 5.66 | 4.26
  Week 8 | 5.66 | 0.00
  Week 12 | 3.77 | 0.00
Statistical Analysis 1: Comparison: CE-224,535 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.121, Barnard exact test; Percent difference = 0.0377, 80% CI 2-sided [-0.00 to 0.09]
Statistical Analysis 2: Comparison: CE-224,535 vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.421, Barnard exact test; Percent difference = 0.0141, 80% CI 2-sided [-0.05 to 0.07]
Statistical Analysis 3: Comparison: CE-224,535 vs Placebo; Week 8: Treatment effect was estimated by the difference of percentages between the treatment groups, and tested using the Barnard exact test; Test type: Superiority or Other; p = 0.058, Barnard exact test; Percent difference = 0.0566, 80% CI 2-sided [0.01 to 0.12]
Statistical Analysis 4: Comparison: CE-224,535 vs Placebo; Week 12: Treatment effect was estimated by the difference of percentages between the treatment groups, and tested using the Barnard exact test; Test type: Superiority or Other; p = 0.121, Barnard exact test; Percent difference = 0.0377, 80% CI 2-sided [-0.00 to 0.09]

5. Secondary Outcome: Number of Tender/Painful and Swollen Joints
Description: Number of tender/painful joints was determined by examining 28 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1. Number of swollen joints was determined by examination of 28 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: FAS included all randomized participants who received at least 1 dose of the randomized study medication. Here, 'number analyzed' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | CE-224,535 | Placebo
Number analyzed (Participants) | 53 | 47
Joints
  Baseline: Tender joints | 13.13 (7.13) | 14.45 (7.03)
  Baseline: Swollen joints | 11.68 (6.30) | 12.45 (6.80)
  Week 2: Tender joints: number analyzed (Participants) | 51 | 47
  Week 2: Tender joints | 10.33 (7.19) | 12.26 (7.11)
  Week 2: Swollen joints: number analyzed (Participants) | 51 | 47
  Week 2: Swollen joints | 8.39 (6.52) | 9.43 (6.45)
  Week 4: Tender joints: number analyzed (Participants) | 47 | 46
  Week 4: Tender joints | 8.64 (6.54) | 10.54 (7.70)
  Week 4: Swollen joints: number analyzed (Participants) | 47 | 46
  Week 4: Swollen joints | 7.47 (6.57) | 7.80 (6.47)
  Week 8: Tender joints: number analyzed (Participants) | 49 | 47
  Week 8: Tender joints | 8.33 (7.35) | 9.81 (6.83)
  Week 8: Swollen joints: number analyzed (Participants) | 49 | 47
  Week 8: Swollen joints | 7.00 (6.16) | 7.57 (6.15)
  Week 12: Tender joints: number analyzed (Participants) | 46 | 40
  Week 12: Tender joints | 7.80 (6.72) | 8.48 (6.89)
  Week 12: Swollen joints: number analyzed (Participants) | 46 | 40
  Week 12: Swollen joints | 6.91 (6.33) | 6.63 (6.23)

6. Secondary Outcome: Physician Global Assessment (PGA) of Arthritis
Description: Physician global assessment of arthritis was measured on a 0 to 100 millimeter (mm) Visual Analog Scale (VAS), with 0 mm= very good and 100 mm= very poor. This was an evaluation based on the participant's disease signs, functional capacity and physical examination.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CE-224,535 | Placebo
Number analyzed (Participants) | 53 | 47
mm
  Baseline | 53.74 (23.82) | 54.83 (23.56)
  Week 2: number analyzed (Participants) | 51 | 46
  Week 2 | 48.04 (25.78) | 50.65 (22.06)
  Week 4: number analyzed (Participants) | 46 | 46
  Week 4 | 42.15 (22.77) | 48.28 (26.22)
  Week 8: number analyzed (Participants) | 49 | 47
  Week 8 | 41.59 (24.87) | 47.72 (25.09)
  Week 12: number analyzed (Participants) | 46 | 40
  Week 12 | 40.02 (25.87) | 41.25 (21.14)

7. Secondary Outcome: Patient's Global Assessment of Arthritis
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 to 100 mm VAS, with 0 mm= very well and 100 mm= very poorly.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CE-224,535 | Placebo
Number analyzed (Participants) | 53 | 47
mm
  Baseline | 56.91 (18.80) | 59.34 (15.19)
  Week 2: number analyzed (Participants) | 51 | 47
  Week 2 | 50.43 (22.24) | 49.66 (21.57)
  Week 4: number analyzed (Participants) | 47 | 46
  Week 4 | 42.94 (20.70) | 42.24 (23.87)
  Week 8: number analyzed (Participants) | 49 | 47
  Week 8 | 43.00 (23.27) | 42.81 (23.68)
  Week 12: number analyzed (Participants) | 46 | 40
  Week 12 | 40.57 (23.26) | 40.00 (21.16)

8. Secondary Outcome: Patient's Global Assessment of Arthritic Pain
Description: Participants measured their pain at the time of assessment on a 0 to 100 mm VAS, with 0 mm= no pain and 100 mm= most severe pain.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: FAS included all randomized participants who received at least 1 dose of the randomized study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'number analyzed' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CE-224,535 | Placebo
Number analyzed (Participants) | 51 | 47
mm
  Baseline: number analyzed (Participants) | 51 | 46
  Baseline | 51.33 (25.08) | 60.13 (20.96)
  Week 2: number analyzed (Participants) | 50 | 47
  Week 2 | 49.20 (23.85) | 51.51 (24.38)
  Week 4: number analyzed (Participants) | 47 | 46
  Week 4 | 43.70 (22.75) | 48.43 (27.20)
  Week 8: number analyzed (Participants) | 49 | 47
  Week 8 | 40.90 (24.94) | 48.79 (24.19)
  Week 12: number analyzed (Participants) | 46 | 40
  Week 12 | 42.07 (27.02) | 43.13 (23.47)

9. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: Health Assessment Questionnaire-Disability Index (HAQ-DI): participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0= no difficulty; 1= some difficulty; 2= much difficulty; 3= unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0= least difficulty and 3= extreme difficulty.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: FAS included all randomized participants who received at least 1 dose of the randomized study medication. Here, 'n' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CE-224,535 | Placebo
Number analyzed (Participants) | 53 | 47
units on a scale
  Baseline | 1.26 (0.68) | 1.38 (0.62)
  Week 2: number analyzed (Participants) | 51 | 47
  Week 2 | 1.15 (0.69) | 1.22 (0.65)
  Week 4: number analyzed (Participants) | 47 | 46
  Week 4 | 1.06 (0.75) | 1.19 (0.74)
  Week 8: number analyzed (Participants) | 49 | 47
  Week 8 | 1.00 (0.75) | 1.23 (0.74)
  Week 12: number analyzed (Participants) | 45 | 40
  Week 12 | 0.97 (0.78) | 1.04 (0.68)

10. Secondary Outcome: Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP])
Description: DAS28-3 (CRP) was calculated from the swollen joint count and tender joint count using the 28 joints count and CRP (milligram per liter [mg/L]). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) less than or equal to (<=) 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-3 (CRP) <2.6 = remission.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CE-224,535 | Placebo
Number analyzed (Participants) | 53 | 47
units on a scale
  Baseline: (n= 53, 47) | 5.11 (0.94) | 5.22 (0.95)
  Week 2: number analyzed (Participants) | 51 | 47
  Week 2 | 4.55 (1.16) | 4.84 (1.12)
  Week 4: number analyzed (Participants) | 45 | 43
  Week 4 | 4.22 (1.32) | 4.48 (1.37)
  Week 8: number analyzed (Participants) | 49 | 46
  Week 8 | 4.21 (1.31) | 4.47 (1.23)
  Week 12: number analyzed (Participants) | 45 | 38
  Week 12 | 4.10 (1.38) | 4.28 (1.22)

11. Secondary Outcome: C-Reactive Protein (CRP)
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | CE-224,535 | Placebo
Number analyzed (Participants) | 53 | 47
milligram per liter (mg/L)
  Baseline | 11.53 (13.78) | 9.22 (9.91)
  Week 2: number analyzed (Participants) | 51 | 47
  Week 2 | 11.04 (14.32) | 9.23 (11.19)
  Week 4: number analyzed (Participants) | 45 | 43
  Week 4 | 11.22 (15.60) | 8.97 (9.29)
  Week 8: number analyzed (Participants) | 49 | 46
  Week 8 | 12.88 (17.96) | 10.38 (12.53)
  Week 12: number analyzed (Participants) | 45 | 38
  Week 12 | 11.85 (17.10) | 9.26 (10.78)

12. Secondary Outcome: Incidence of Withdrawal Due to Lack of Efficacy
Description: Number of participants who withrew due to lack of efficacy were reported.
Time Frame: Week 2, 4, 8, 12, 14
Population: FAS included all randomized participants who received at least 1 dose of the randomized study medication.
Measure: Number; unit: participants
Arm/Group | CE-224,535 | Placebo
Number analyzed (Participants) | 53 | 47
participants
  Week 2 | 0 | 0
  Week 4 | 0 | 0
  Week 8 | 0 | 0
  Week 12 | 0 | 3
  Week 14 | 0 | 3
Statistical Analysis 1: Comparison: CE-224,535 vs Placebo; Week 2: p-value was analyzed using Barnard Exact Test; Test type: Superiority or Other; p = 1.0000, Barnard exact test
Statistical Analysis 2: Comparison: CE-224,535 vs Placebo; Week 4: p-value was analyzed using Barnard Exact Test; Test type: Superiority or Other; p = 1.0000, Barnard exact test
Statistical Analysis 3: Comparison: CE-224,535 vs Placebo; Week 8: p-value was analyzed using Barnard Exact Test; Test type: Superiority or Other; p = 1.0000, Barnard exact test
Statistical Analysis 4: Comparison: CE-224,535 vs Placebo; Week 12: p-value was analyzed using Barnard Exact Test; Test type: Superiority or Other; p = 0.0637, Barnard exact test
Statistical Analysis 5: Comparison: CE-224,535 vs Placebo; Week 14: p-value was analyzed using Barnard Exact Test; Test type: Superiority or Other; p = 0.0637, Barnard exact test

13. Secondary Outcome: Time to Withdrawal Due to Lack of Efficacy
Time Frame: Baseline up to Week 14
Population: Results are not reported because median time could not be estimated as very few participants discontinued study due to lack of efficacy.
Groups:
- CE-224,535: CE-224,535 500 milligram (mg) tablet twice daily for 12 weeks.
- Placebo: Placebo matched to CE-224,535 500 milligram (mg) tablet twice daily for 12 weeks.
Arm/Group | CE-224,535 | Placebo
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: CE-224,535 Plasma Concentrations
Description: Nominal times were used for summarizing the pharmacokinetic results (0 hours at randomization [Day 1] and Week 4 [pre-dose]; 1 hour at Week 2 [post-dose]; 2 hours at randomization [post-dose on Day 1]; and 3 hours at Week 2 [post-dose] and Week 4 [post-dose]).
Time Frame: 0 hour (pre-dose), 2 hours post-dose at Day 1; 1, 3 hours post-dose at Week 2; 0 hour (pre-dose), 3 hours post-dose at Week 4
Population: FAS included all randomized participants who received at least 1 dose of the randomized study medication.
Measure: Median (Full Range); unit: nanogram per milliliter (ng/mL)
Arm/Group | CE-224,535
Number analyzed (Participants) | 53
nanogram per milliliter (ng/mL)
  0 hour | 256 [13 to 4060]
  1 hour | 3110 [56 to 8690]
  2 hours | 4280 [1170 to 10200]
  3 hours | 2935 [90 to 11500]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CE-224,535 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/53 | 1/47
Other Adverse Events (participants affected / at risk) | 32/53 | 26/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CE-224,535 (N=53) | Placebo (N=47)
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Capsular contracture associated with breast implant (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Breast prosthesis implantation (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CE-224,535 (N=53) | Placebo (N=47)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ear canal erythema (Ear and labyrinth disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Eructation (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 2
Oral disorder (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1
Fatigue (General disorders) | 1 | 0
Feeling hot (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 3 | 1
Folliculitis (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 3 | 1
Oral herpes (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Viral infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 | 2
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 3 | 4
Lethargy (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 3
Renal failure (Renal and urinary disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.